CLINICAL TRIAL: NCT02610335
Title: Evaluation of Spinal Mobility Reeducation in Patients Treated for a Lumbar Spinal Stenosis After Epidural Infiltration. Randomized and Comparative Study: Kyphosis Reeducation Versus Spinal Mobility Reeducation
Brief Title: Evaluation of Spinal Mobility Reeducation in Patients Treated for a Lumbar Spinal Stenosis After Epidural Infiltration
Acronym: CLEMOB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment of participants was very difficult despite a change in the organisation. The inclusion criteria did not result in the expected number of participants, and the credits ran out.
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2012/36
Record Dates: First submitted 2015-06-04; First posted 2015-11-20 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Lumbar Spinal Stenosis
Keywords: lumbar spinal stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (C) (Active Comparator): Kyphosis reeducation + patient education + auto-reeducation at home
  Interventions: Other: Control group (C)
- Test group (M) (Other): Spinal mobility reeducation + patient education + auto-reeducation at home.
  Interventions: Other: Test group

INTERVENTIONS:
Other: Control group (C) — * kyphosis reeducation on Huber platform during 2 weeks,
  * patient education : on physiopathology of the lumbar spinal stenosis and treatments as well as healthy lifestyle and prevention (plans of anatomy, plastic column, slides of medical imaging),
  * flexibility exercises, stretching exercises and abdominal muscles exercises : to continue at home (the exercises will be reported on a book that will be given to the patient),
  * exercises on cycle ergometer or walking on treadmill : to continue at home.
  Arms: Control group (C)
Other: Test group — * spinal mobility reeducation on Huber platform during 2 weeks,
  * patient education : on physiopathology of the lumbar spinal stenosis and treatments as well as healthy lifestyle and prevention (plans of anatomy, plastic column, slides of medical imaging),
  * flexibility exercises and mobilization exercises : to continue at home (the exercises will be reported on a book that will be given to the patient),
  * exercises on cycle ergometer or walking on treadmill : to continue at home.
  Arms: Test group (M)

SUMMARY:
In actual practice the patients with mild or moderate lumbar spinal stenosis symptoms receive an epidural infiltration and participate in kyphosis reeducation in first intention. Yet the kyphosis reeducation did not show a real profit in the time compared with the natural evolution of the pathology. The study assume that the spinal mobility reeducation will reduce the incidence of pain recurrences compared with the classic kyphosis reeducation.

DETAILED DESCRIPTION:
The standard treatment of lumbar spinal stenosis is the lumbar canal recalibration surgery which presents co-morbidity factors and risks of post-operative complications. The non-invasive methods are a good alternative compared with the surgery : the patients medically treated present few damages and the results of the postponed surgery are equivalent to the immediate surgery. That is why a non-surgical treatment is proposed in first intention to the patients with mild or moderate symptoms : this treatment associates an epidural infiltration and a kyphosis reeducation.

Yet the kyphosis reeducation did not show a real profit in the time compared with the natural evolution of the pathology. The benefits of the infiltration are lost three months after this one in 80 % of the cases. A return to physical activity and a restored spinal mobility would improve the duration of the infiltration effect. The objective is then to compare the efficiency of a spinal mobility reeducation program versus a kyphosis reeducation program in patients with acquired and central lumbar spinal stenosis. It is a prospective, monocentric, randomized, superiority and parallel-group study :

* group C (control group) : kyphosis reeducation + patient education + auto-reeducation at home,
* group M (test group) : spinal mobility reeducation + patient education + auto-reeducation at home.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years,
* central, acquired and multi-staged lumbar spinal stenosis,
* pain since at least three months,
* radicular pains higher than the lumbar pains,
* walking distance < 1000 m,
* oral consent.

Exclusion Criteria:

* intercurrent pathology limiting the walking distance (arteriopathy, cardio-respiratory insufficiency, disabling arthrosis affecting the lower limbs...),
* history of spinal surgery for lumbar spinal stenosis,
* extended lumbar arthrodesis (equal to or greater than 2 levels),
* monosegmental and degenerative spondylolisthesis,
* foraminal stenosis,
* motor deficit of the lower limbs or Cauda equina syndrome ("Cauda equina" syndrome (CES) is a serious neurologic condition in which damage to the cauda equina causes acute loss of function of the lumbar plexus, (nerve roots) of the spinal canal below the termination (conus medullaris) of the spinal cord),
* bleeding disorders or allergies contraindicating the epidural infiltration.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
maximal walking distance | the 90 days visit
  : ratio between the maximal walking distance at the 90 days visit and the maximal walking distance at the Day 4 in percent. Walking on a plane road, 70 m in length, without obstacle and with markings every 10 meters (total length : not more than 2 km).

SECONDARY OUTCOMES:
evaluation of the lumbar pain | Day 0
  evaluation of the lumbar pain: measured by a verbal analog scale 0-100 mm (0 : no pain, 100 : maximal pain),
evaluation of the lumbar pain | Day 4
  evaluation of the lumbar pain: measured by a verbal analog scale 0-100 mm (0 : no pain, 100 : maximal pain),
evaluation of the lumbar pain | Day 30
  evaluation of the lumbar pain: measured by a verbal analog scale 0-100 mm (0 : no pain, 100 : maximal pain),
evaluation of the lumbar pain | Day 90
  evaluation of the lumbar pain: measured by a verbal analog scale 0-100 mm (0 : no pain, 100 : maximal pain),
evaluation of the lumbar pain | Day 365
  evaluation of the lumbar pain: measured by a verbal analog scale 0-100 mm (0 : no pain, 100 : maximal pain),
evaluation of the radicular pain | Day 0
  measured by a verbal analog scale 0-100 mm (0 : no pain, 100 : maximal pain),
evaluation of the radicular pain | Day 4
  measured by a verbal analog scale 0-100 mm (0 : no pain, 100 : maximal pain),
evaluation of the radicular pain | Day 30
  measured by a verbal analog scale 0-100 mm (0 : no pain, 100 : maximal pain),
evaluation of the radicular pain | Day 90
  measured by a verbal analog scale 0-100 mm (0 : no pain, 100 : maximal pain),
evaluation of the radicular pain | Day 365
  measured by a verbal analog scale 0-100 mm (0 : no pain, 100 : maximal pain),
evaluation scales | Day 0
  evaluation scales : score of Quebec (functional impotence)
evaluation scales | Day 4
  evaluation scales : score of Quebec (functional impotence)
evaluation scales | Day 30
  evaluation scales : score of Quebec (functional impotence)
evaluation scales | Day 90
  evaluation scales : score of Quebec (functional impotence)
evaluation scales | Day 365
  evaluation scales : score of Quebec (functional impotence)
maximal walking distance | Day 0
  maximal walking distance : on a defined road
maximal walking distance | Day 4
  maximal walking distance : on a defined road
maximal walking distance | Day 30
  maximal walking distance : on a defined road
maximal walking distance | Day 90
  maximal walking distance : on a defined road
maximal walking distance | Day 365
  maximal walking distance : on a defined road
compliance with the auto-reeducation at home | Day 30
  compliance with the auto-reeducation at home : questionnaire.
compliance with the auto-reeducation at home | Day 90
  compliance with the auto-reeducation at home : questionnaire.
compliance with the auto-reeducation at home | Day 365
  compliance with the auto-reeducation at home : questionnaire.
Score of Japanese Orthopaedic Association (llumbar radiculopathy) | Day 4
Score of Japanese Orthopaedic Association (llumbar radiculopathy) | Day 30
Score of Japanese Orthopaedic Association (llumbar radiculopathy) | Day 90
Score of Japanese Orthopaedic Association (llumbar radiculopathy) | Day 365
score of "Douleur Neuropathique 4" (DN4 - neuropathy) | Day 4
score of "Douleur Neuropathique 4" (DN4 - neuropathy) | Day 30
score of "Douleur Neuropathique 4" (DN4 - neuropathy) | Day 90
score of "Douleur Neuropathique 4" (DN4 - neuropathy) | Day 365
score Medical Outcomes Study Short-Form General Health Survey 12 (health status) | Day 4
score Medical Outcomes Study Short-Form General Health Survey 12 (health status) | Day 30
score Medical Outcomes Study Short-Form General Health Survey 12 (health status) | Day 90
score Medical Outcomes Study Short-Form General Health Survey 12 (health status) | Day 365

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu DE-SÈZE, MD, Study Director — service de médecine physique et de réadaptation, Centre Hospitalier Universitaire de Bordeaux,; Antoine BENARD, MD, Study Chair — USMR CHU Bordeaux
Locations (1):
- University Hospital of Bordeaux - Hospital Pellegrin, Bordeaux, France

REFERENCES:
- [Background] Berney J. [Epidemiology of narrow spinal canal]. Neurochirurgie. 1994;40(3):174-8. French. PMID 7723924
- [Background] Weinstein JN, Lurie JD, Tosteson TD, Hanscom B, Tosteson AN, Blood EA, Birkmeyer NJ, Hilibrand AS, Herkowitz H, Cammisa FP, Albert TJ, Emery SE, Lenke LG, Abdu WA, Longley M, Errico TJ, Hu SS. Surgical versus nonsurgical treatment for lumbar degenerative spondylolisthesis. N Engl J Med. 2007 May 31;356(22):2257-70. doi: 10.1056/NEJMoa070302. PMID 17538085
- [Background] Yamashita K, Ohzono K, Hiroshima K. Five-year outcomes of surgical treatment for degenerative lumbar spinal stenosis: a prospective observational study of symptom severity at standard intervals after surgery. Spine (Phila Pa 1976). 2006 Jun 1;31(13):1484-90. doi: 10.1097/01.brs.0000219940.26390.26. PMID 16741459
- [Background] Rillardon L, Guigui P, Veil-Picard A, Slulittel H, Deburge A. [Long-term results of surgical treatment of lumbar spinal stenosis]. Rev Chir Orthop Reparatrice Appar Mot. 2003 Nov;89(7):621-31. French. PMID 14699308
- [Background] Lieberman I. Surgery reduced pain and disability in lumbar spinal stenosis better than nonoperative treatment. J Bone Joint Surg Am. 2007 Aug;89(8):1872. doi: 10.2106/JBJS.8908.ebo2. No abstract available. PMID 17671033